CLINICAL TRIAL: NCT02545712
Title: Safe Excipient Exposure in Neonates and Small ChildreN - a Retrospective, Descriptive Study Off the Amount of Ethanol, Propylene Glycol, Benzyl Alcohol, Parabens, Acesulfam k, Aspartame, Glycerol, Sorbitol and Polysorbate-80 Exposed to Pediatric Patients
Brief Title: Safe Excipient Exposure in Neonates and Small ChildreN
Acronym: SEEN
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Bispebjerg Hospital (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Kristine Svinning Valeur, MS, Bispebjerg Hospital
Other Study IDs: BBH-KSV-01
Record Dates: First submitted 2015-09-03; First posted 2015-09-10 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Excipient Exposure; Neonatal; Pediatric
Keywords: Ethanol; Propylene glycol; Benzyl alcohol; Acesulfam potassium; Aspartame; Glycerin; Sorbitol; Methyl-p-hydroxybenzoate; Propanyl-p-hydroxybenzoate; Patients
MeSH Terms: interventions — Ethanol; acetosulfame; Glycerol

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Neonatal patients: Receiving 2 or more drugs at one day during their hospitalisation. For each drug, it is listed whether it is an extemporaneous, registered, the preparation, dosis, amount, interval, formulation and route of administration. It is noted if the drug contains ethanol, propylene glycol, benzyl alcohol, methyl-p-hydroxybenzoate, propanyl-p-hydroxybenzoate, acesulfam potassium, aspartame, glycerin and/or sorbitol.
  Interventions: Other: Exposure to ethanol; Other: Exposure to propylene glycol; Other: Exposure to benzyl alcohol; Other: Exposure to acesulfam potassium; Other: Exposure to aspartame; Other: Exposure to glycerol; Other: Exposure to sorbitol; Other: Exposure to methyl-p-hydroxybenzoate; Other: Exposure to propanyl-p-hydroxybenzoate; Other: Exposure to polysorbate-80
- Pediatric patients (28 days ≤ 5 years): Receiving 3 or more drugs at one day during their hospitalisation. For each drug, it is listed whether it is an extemporaneous, registered, the preparation, dosis, amount, interval, formulation and route of administration. It is noted if the drug contains ethanol, propylene glycol, benzyl alcohol, methyl-p-hydroxybenzoate, propanyl-p-hydroxybenzoate, acesulfam potassium, aspartame, glycerin and/or sorbitol.
  Interventions: Other: Exposure to ethanol; Other: Exposure to propylene glycol; Other: Exposure to benzyl alcohol; Other: Exposure to acesulfam potassium; Other: Exposure to aspartame; Other: Exposure to glycerol; Other: Exposure to sorbitol; Other: Exposure to methyl-p-hydroxybenzoate; Other: Exposure to propanyl-p-hydroxybenzoate; Other: Exposure to polysorbate-80

INTERVENTIONS:
Other: Exposure to ethanol — The drug source(s) and amount administered daily are noted.
  Other Names: Ethyl achohol
Other: Exposure to propylene glycol — The drug source(s) and amount administered daily are noted.
Other: Exposure to benzyl alcohol — The drug source(s) and amount administered daily are noted.
Other: Exposure to acesulfam potassium — The drug source(s) and amount administered daily are noted.
  Other Names: Acesulfame-K
Other: Exposure to aspartame — The drug source(s) and amount administered daily are noted.
Other: Exposure to glycerol — The drug source(s) and amount administered daily are noted.
  Other Names: Glycerol
Other: Exposure to sorbitol — The drug source(s) and amount administered daily are noted.
Other: Exposure to methyl-p-hydroxybenzoate — The drug source(s) and amount administered daily are noted.
  Other Names: including sodium-methyl-p-hydroxybenzoate
Other: Exposure to propanyl-p-hydroxybenzoate — The drug source(s) and amount administered daily are noted.
  Other Names: including sodium-propanyl-p-hydroxybenzoate
Other: Exposure to polysorbate-80 — The drug source(s) and amount administered daily are noted.

SUMMARY:
The purpose of this study is to explore the quantity of excipient exposure in neonatal and young pediatric patients in a Danish Hospital. The focus will be on the preservatives ethanol, propyl glycol, benzyl alcohol, methyl-p-hydroxybenzoate and propanyl-p-hydroxybenzoate and the artificial sweeteners acesulfam potassium, aspartame, glycerol and sorbitol.

DETAILED DESCRIPTION:
Studies have previously examined whether or not neonatal nor pediatric patients are exposed to excipients and what excipients they are possibly exposed to. They have shown that practically all neonatal patients receive one or more drug containing an excipient, known to be harmful. This observational study will look at both registered drugs and extemporaneous pharmaceuticals as possible sources of excipients. Based on information provided by the manufacturer (ex. the index-list), the investigator will calculate the amounts of excipients administered to the patient a week after hospitalisation. The investigator will calculate the blood alcohol content when the neonatal patient are exposed to ethanol and/or propylene glycol.

By grouping the patients according to age and subgrouping according to diagnosis/affected organ system and compare the amount of excipient exposure in each group, the study aims at identifying the most vulnerable neonatal and/or pediatric patients in terms of the amount and identity of excipients accumulated in the patient.

The study will use a descriptive, parametric statistic analysis to identify

* an average exposure rate (concentration i mg/l or amount in mg) of each of the listed excipients
* how much the average patient in each age-group is exposed to each excipient
* how much the average patient in each "affected organ system"-subgroup is exposed to each excipient

ELIGIBILITY:
Inclusion Criteria:

* if < 28 days: must receive 2 or more prescriptions a day
* if 28 days ≤ 5 years: must receive 3 or more prescriptions a day
* must have been/be submitted and treated at the neonatal department (units 5021, 5023, 5024) or pediatric department (units 5061, 5062, 5054, 4144) of Rigshospitalet

Exclusion Criteria:

* no up-dated weight is listed
* > 5 years old

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonatal patients and pediatric patients (≤ 5 years) who, at one point, have been/are being treated at the "Neonatalklinikken" (units 5021, 5023, 5024) or "BørneUngeklinikken" (units 5061, 5062, 5054, 4144) of Rigshospitalet, Denmark. To be included in the study, the patients must receive
  * 2 or more different drugs if < 28 days old
  * 3 or more different drugs if 28 day ≤ 5 years old
Sampling Method: Non-Probability Sample
Enrollment: 630 (Actual)
Dates: Start 2016-01; Primary Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Blood alcohol content measured in per mille (grams of ethanol and propylene glycol pr. kilograms of blood) in the patient | Single day
  Both concentrations of ethanol and propylene glycol are included in the calculations. with propylene glycol 1/3 as intoxicating as ethanol.
Concentration (mg/kg/day) of benzyl alcohol in the patient | Single day
Concentration (mg/kg/day) of acesulfam potassium in the patient | Single day
Concentration (mg/kg/day) of aspartame in the patient | Single day
Concentration (mg/kg/day) of glycerin in the patient | Single day
Concentration (mg/kg/day) of sorbitol in the patient | Single day
Concentration (mg/l) of methyl-p-hydroxybenzoate in the patient | Single day
Concentration (mg/kg/day) of propyl-p-hydroxybenzoate in the patient | Single day
Concentration (mg/kg/day) of polysorbate-80 in the patient | Single day

SECONDARY OUTCOMES:
Identification of patient group (according to age-interval) most vulnerable to excipient exposure (measured in number of excipients) | During the participants hospitalization, an expected average of 2 months
  The excipients (ethanol, propylene glycol, benzyl alcohol, methyl-p-hydroxybenzoate, propyl-p-hydroxybenzoate, acesulfam potassium, aspartame, glycerol, polysorbate-80 and sorbitol) will be ranked according to which excipient is most often present in the medicine administered to the patients.
Identification of patient group (according to age-interval) most vulnerable to excipient exposure (amounts of each excipient measured in (mg/l)) | During the participants hospitalization, an expected average of 2 months
  The excipients (ethanol, propylene glycol, benzyl alcohol, methyl-p-hydroxybenzoate, propyl-p-hydroxybenzoate, acesulfam potassium, aspartame, glycerol, polysorbate-80 and sorbitol) will be ranked according to which excipient is most often present in the medicine administered to the patients.
Identification of patient group (according to affected organ system) most vulnerable to excipient exposure (measured in number of excipients) | During the participants hospitalization, an expected average of 2 months
  The excipients (ethanol, propylene glycol, benzyl alcohol, methyl-p-hydroxybenzoate, propyl-p-hydroxybenzoate, acesulfam potassium, aspartame, glycerol, polysorbate-80 and sorbitol) will be ranked according to which excipient is most often present in the medicine administered to the patients.
Identification of patient group (according to affected organ system) most vulnerable to excipient exposure (amounts of each excipient measured in (mg/l)) | During the participants hospitalization, an expected average of 2 months
  The excipients (ethanol, propylene glycol, benzyl alcohol, methyl-p-hydroxybenzoate, propyl-p-hydroxybenzoate, acesulfam potassium, aspartame, glycerol, polysorbate-80 and sorbitol) will be ranked according to which excipient is most often present in the medicine administered to the patients.
Identification of number of patient exposed to ethanol levels above tolerance levels proposed by international medicines agencies like EMA and FDA | Single day
  Comparison of each patient daily exposure rate of ethanol to daily tolerance limit
Identification of number of patient exposed to propylene glycol levels above tolerance levels proposed by international medicines agencies like EMA and FDA | Single day
  Comparison of each patient daily exposure rate of proplyene glycol to daily tolerance limit
Identification of number of patient exposed to benzyl alcohol levels above tolerance levels proposed by international medicines agencies like EMA and FDA | Single day
  Comparison of each patient daily exposure rate of benzyl alcohol to daily tolerance limit
Identification of number of patient exposed to methyl-p-hydroxy-benzoate levels above tolerance levels proposed by international medicines agencies like EMA and FDA | Single day
  Comparison of each patient daily exposure rate of methyl-p-hydroxy-benzoate to daily tolerance limit
Identification of number of patient exposed to propyl-p-hydroxy-benzoate levels above tolerance levels proposed by international medicines agencies like EMA and FDA | Single day
  Comparison of each patient daily exposure rate of propyl-p-hydroxy-benzoate to daily tolerance limit
Identification of number of patient exposed to sodium-propyl-p-hydroxy-benzoate levels above tolerance levels proposed by international medicines agencies like EMA and FDA | Single day
  Comparison of each patient daily exposure rate of sodium-propyl-p-hydroxy-benzoate to daily tolerance limit
Identification of number of patient exposed to sodium-methyl-p-hydroxy-benzoate levels above tolerance levels proposed by international medicines agencies like EMA and FDA | Single day
  Comparison of each patient daily exposure rate of sodium-methyl-p-hydroxy-benzoate to daily tolerance limit
Identification of number of patient exposed to acesulfame potassium levels above tolerance levels proposed by international medicines agencies like EMA and FDA | Single day
  Comparison of each patient daily exposure rate of acesulfame potassium to daily tolerance limit
Identification of number of patient exposed to aspartame levels above tolerance levels proposed by international medicines agencies like EMA and FDA | Single day
  Comparison of each patient daily exposure rate of aspartame to daily tolerance limit
Identification of number of patient exposed to glycerol levels above tolerance levels proposed by international medicines agencies like EMA and FDA | Single day
  Comparison of each patient daily exposure rate of glycerol to daily tolerance limit
Identification of number of patient exposed to sorbitol levels above tolerance levels proposed by international medicines agencies like EMA and FDA | Single day
  Comparison of each patient daily exposure rate of sorbitol to daily tolerance limit
Identification of number of patient exposed to polysorbate-80 levels above tolerance levels proposed by international medicines agencies like EMA and FDA | Single day
  Comparison of each patient daily exposure rate of polysorbate-80 to daily tolerance limit

CONTACTS AND LOCATIONS:
Overall Officials: Kristine Svinning Valeur, MS, Principal Investigator — University Hospital Bispebjerg and Frederiksberg

REFERENCES:
- [Background] Nellis G, Metsvaht T, Varendi H, Toompere K, Lass J, Mesek I, Nunn AJ, Turner MA, Lutsar I; ESNEE consortium. Potentially harmful excipients in neonatal medicines: a pan-European observational study. Arch Dis Child. 2015 Jul;100(7):694-9. doi: 10.1136/archdischild-2014-307793. Epub 2015 Apr 8. PMID 25854872
- [Background] Souza A Jr, Santos D, Fonseca S, Medeiros M, Batista L, Turner M, Coelho H. Toxic excipients in medications for neonates in Brazil. Eur J Pediatr. 2014 Jul;173(7):935-45. doi: 10.1007/s00431-014-2272-z. Epub 2014 Feb 6. PMID 24500397
- [Background] Marek E, Kraft WK. Ethanol pharmacokinetics in neonates and infants. Curr Ther Res Clin Exp. 2014 Oct 22;76:90-7. doi: 10.1016/j.curtheres.2014.09.002. eCollection 2014 Dec. PMID 25379066
- [Background] Nguyen KA, Claris O, Kassai B. Unlicensed and off-label drug use in a neonatal unit in France. Acta Paediatr. 2011 Apr;100(4):615-7. doi: 10.1111/j.1651-2227.2010.02103.x. Epub 2010 Dec 17. No abstract available. PMID 21410525
- [Background] Jacqz-Aigrain E. Drug policy in Europe Research and funding in neonates: current challenges, future perspectives, new opportunities. Early Hum Dev. 2011 Mar;87 Suppl 1:S27-30. doi: 10.1016/j.earlhumdev.2011.01.007. Epub 2011 Jan 26. PMID 21269785
- [Background] Allegaert K. Neonates need tailored drug formulations. World J Clin Pediatr. 2013 Feb 8;2(1):1-5. doi: 10.5409/wjcp.v2.i1.1. eCollection 2013 Feb 8. PMID 25254168
- [Background] Bellis JR, Kirkham JJ, Thiesen S, Conroy EJ, Bracken LE, Mannix HL, Bird KA, Duncan JC, Peak M, Turner MA, Smyth RL, Nunn AJ, Pirmohamed M. Adverse drug reactions and off-label and unlicensed medicines in children: a nested case-control study of inpatients in a pediatric hospital. BMC Med. 2013 Nov 7;11:238. doi: 10.1186/1741-7015-11-238. PMID 24229060
- [Background] Nahata MC. Safety of "inert" additives or excipients in paediatric medicines. Arch Dis Child Fetal Neonatal Ed. 2009 Nov;94(6):F392-3. doi: 10.1136/adc.2009.160192. No abstract available. PMID 19846397
- [Background] Whittaker A, Currie AE, Turner MA, Field DJ, Mulla H, Pandya HC. Toxic additives in medication for preterm infants. Arch Dis Child Fetal Neonatal Ed. 2009 Jul;94(4):F236-40. doi: 10.1136/adc.2008.146035. Epub 2009 Jan 21. PMID 19158148
- [Background] Saiyed MM, Lalwani T, Rana D. Is off-label use a risk factor for adverse drug reactions in pediatric patients? A prospective study in an Indian tertiary care hospital. Int J Risk Saf Med. 2015;27(1):45-53. doi: 10.3233/JRS-150642. PMID 25766066
- [Background] Collison KS, Makhoul NJ, Zaidi MZ, Al-Rabiah R, Inglis A, Andres BL, Ubungen R, Shoukri M, Al-Mohanna FA. Interactive effects of neonatal exposure to monosodium glutamate and aspartame on glucose homeostasis. Nutr Metab (Lond). 2012 Jun 14;9(1):58. doi: 10.1186/1743-7075-9-58. PMID 22697049
- [Background] Ornoy A, Ergaz Z. Alcohol abuse in pregnant women: effects on the fetus and newborn, mode of action and maternal treatment. Int J Environ Res Public Health. 2010 Feb;7(2):364-79. doi: 10.3390/ijerph7020364. Epub 2010 Jan 27. PMID 20616979
- [Background] Lass J, Kaar R, Jogi K, Varendi H, Metsvaht T, Lutsar I. Drug utilisation pattern and off-label use of medicines in Estonian neonatal units. Eur J Clin Pharmacol. 2011 Dec;67(12):1263-71. doi: 10.1007/s00228-011-1072-x. Epub 2011 Jun 11. PMID 21667125
- [Background] Fister P, Urh S, Karner A, Krzan M, Paro-Panjan D. The prevalence and pattern of pharmaceutical and excipient exposure in a neonatal unit in Slovenia. J Matern Fetal Neonatal Med. 2015;28(17):2053-61. doi: 10.3109/14767058.2014.976549. Epub 2015 Sep 4. PMID 25316561
- [Derived] Valeur KS, Hertel SA, Lundstrom KE, Holst H. Safe excipient exposure in neonates and small children - protocol for the SEEN project. Dan Med J. 2017 Feb;64(2):A5324. PMID 28157063
- See also: Isaac R, Khan I, Langley C. Ethanol intake of paediatric intensive care patients. Arch Dis Child 2013;98:e1 doi:10.1136/archdischild-2013-303935a.21 — http://adc.bmj.com/content/98/6/e1.14.short